CLINICAL TRIAL: NCT03414138
Title: Identifying the Neurofunctional Connections Supporting Mindfulness Meditation Based Analgesia
Brief Title: Brain Mechanisms Supporting Meditation-based Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Fadel Zeidan, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00040373; 4R00AT008238-03 (NIH)
Record Dates: First submitted 2018-01-16; First posted 2018-01-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: Pain; Mindfulness; Meditation; fMRI
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Healthy research participants, trained to psychophysically rate their experience in response to a range of thermal stimuli, will be randomly assigned to one of two experimental groups (mindfulness meditation n=20 or deep-breathing meditation n=20). After receiving four twenty-minute meditation training sessions, participants will return for a final session of thermal testing while lying in the MRI scanner. Participants will be exposed to 4 blocks of testing, using thermal stimuli cycled between painful (49°C) and non-painful (35°C) temperatures for 6 minutes. Blood oxygen-level dependent imaging will be used to map the functional connectivity of brain regions in response to the thermal fluctuations. In the first two blocks participants will lie quietly with eyes closed. After a 10 minute rest, subjects will begin meditating and the thermal testing will resume.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomly assigned to two groups by the research coordinator. Investigators, study staff and MRI technicians will be blind as to the participant's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation Group (Experimental): Research volunteers will participate in four sessions (20 min/session) of mindfulness training. Participants are taught that perceived sensory events are "momentary" and "fleeting", requiring no further evaluation. They will be asked to close their eyes, relax and focus on the flow of their breathing by "simply letting go" of discursive thoughts.
  Interventions: Behavioral: Mindfulness Training
- Book Listening Control (Active Comparator): Study volunteers will listen to an audio recording of the Natural History of Selborne across each session.This 4 session sequence is meant to match features of the experimental meditation sessions, including attention to the recording, room setting, social support, conditioning, and time elapsed during the sessions. We do not expect that this group will demonstrate significant blood oxygenation changes as a function of the intervention.
  Interventions: Behavioral: Book Listening Control

INTERVENTIONS:
Behavioral: Mindfulness Training — A well-validated brief mindfulness-based mental training regimen [four sessions; 20 min/session] will be used to teach patients to independently practice mindfulness meditation.
  Other Names: mental training
  Arms: Mindfulness Meditation Group
Behavioral: Book Listening Control — Study volunteers will listen to four 20 minute blocks of The Natural History and Antiquities of Selborne throughout their interventions.
  Other Names: mental training
  Arms: Book Listening Control

SUMMARY:
Mindfulness meditation has been shown to reduce pain in experimental and clinical settings, and the neural mechanisms underlying this analgesia are distinct from that of placebo related beliefs in the utility of the meditation. Although previous studies have identified potential cortical and sub-cortical targets responsible for mediating these effects, the connectional relationships between them remains largely unexplored. The present study will use blood-oxygen-level dependent (BOLD) neuroimaging to assess functional connections supporting mindfulness meditation.

DETAILED DESCRIPTION:
Mindfulness meditation, significantly reduces pain in experimental and clinical settings. Although findings from this laboratory provide novel insights into some of the brain mechanisms supporting the modulation of pain by meditation , the specific analgesic mechanisms engaged during mindfulness meditation remain poorly characterized.

To date, there are no studies that have identified the neurofunctional connections supporting mindfulness meditation-based pain relief. Employing fMRI, the objective of this study will be to determine the neural systems of action supporting mindfulness-based pain relief. The study will determine if higher order brain regions are involved in mindfulness-based analgesia. The results from this aim will identify a neural marker(s) for meditation-related pain relief, a critical step in defining how meditation reduces pain.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers between ages 18 and 65.
* Men and women of all races will be included

Exclusion Criteria:

* Subjects with a history of psychiatric or neurological disorders.
* Subjects will be excluded if they report being claustrophobic.
* Subjects with a prior history of meditation training will be excluded.
* Subjects with ferrous metal or electronic devices (e g., pacemakers) implanted in there body will be excluded.
* Pregnant subjects will be excluded.
* Subjects that demonstrate no pain to noxious temperatures (>49°C) or excessive responses to temperatures at or below 43°C will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) signaling | Up to 3 weeks
  Changes in blood oxygenation levels to thermally noxious stimuli (49°C) will be assessed, and planned comparisons will be performed between subjects trained in mindfulness meditation and those trained in deep-breathing meditation.

SECONDARY OUTCOMES:
Change in Visual Analog Scale Pain Ratings as a function of mindfulness-based mental training | Up to 3 weeks
  The visual analog scale (VAS) measures pain ratings that will be assessed in response to noxious (49°C) thermal stimuli applied to the back of the right calf muscle.
  Pain intensity and pain unpleasantness ratings will be assessed with a Visual Analog Scale. The minimum rating ("0") is designated as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable". Higher values corresponded to higher perceived pain ratings.
  Baseline pain ratings will be assessed on session one and again at session six.

OTHER OUTCOMES:
Respiration Rate | Up to 3 weeks
  A respiratory transducer (TSD 201; Biopac Systems) will be placed around the chest to measure the paticipant's rate of respiration.
Heart Rate | up to 3 weeks
  Pulse oximeter (OXY-MRI-SPO2; Biopac Systems) will be placed on the left index finger to measure the paticipant's heart rate.
State Anxiety Inventory (SAI) | up to 3 weeks
  This inventory is a 20 question test used to measure a subject's state of anxiety. A numeric value between 1 (Not at all) and 4 (Very Much So) is provided in response to each statement. The range of scores for this test is between 20 and 80, with higher scores reflecting higher estimates of anxiety.
Freiburg Mindfulness Inventory (FMI) | up to 3 weeks
  The FMI is a 14 item measure of mindfulness. Each declarative statement is measured on a 4 point scale ranging from: 1 (Rarely) to 4 (Almost Always). A couple of the items are reverse scored. Higher scores reflect higher states of mindfulness.
Beck's Depression Inventory (BDI) | up to 3 weeks
  This a 21-item multiple choice self-report inventory used to measure the severity of depression. A score between 0 and 3 is applied to each question. Higher total scores indicate more severe depressive symptoms.
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression
Multidimensional Iowa Suggestibility Scale (MISS) short form | up to 3 weeks
  The MISS includes five suggestibility subscales (consumer, physiological, physiological reactivity, persuadability, and peer conformity) and two companion scales (unpersuadability and the short suggestibility scale). The five suggestibility subscales can be summed to give the suggestibility total score. Higher values equate to higher levels of suggestibility.
Positive and Negative Affective Scale (PANAS) | up to 3 weeks
  PANAS is composed of two mood scales, one that measures positive affect and the other which measures negative affect. It uses a 20 item test that employs a 5-point rating scale ranging from very slightly or not at all (1) to extremely so (5). Positive affect scores and negative affect scores are calculated separately by adding each group independently. For the positive items, higher scores represent higher levels of positive affect. For the negative items, lower scores represent lower levels of negative affect.
Attitude Toward Treatment Inventory (ATTI) | up to 3 weeks
  The ATTI is used to monitor a participant's impressions and attitudes about the interventions used in this study (i.e. mindfulness meditation). It supplies 5 multiple-choice questions answered on a 10 point scale, ranging from 0 (not logical) to 9 (very logical). Higher scores reflect more positive subject impressions about the therapeutic interventions.
Pain Catastrophizing Scale (PCS) | up to 3 weeks
  The PCS is a 13 item scale, with each item rated on a 5-point scale between: 0 (Not at all) and 4 (all the time). The PCS is broken into three subscales including: magnification, rumination, and helplessness. The total range of scores is between 0-52 with higher values reflecting more salient impacts of pain on one's day to day experience.
Profile of Mood States (PoMS) Questionnaire | up to 3 weeks
  The PoMS is a psychological rating scale used to assess transient and distinct mood states. The POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A five-point scale ranging from "not at all" (0) to "extremely" (4) is provided for participants to rate their mood to 65 descriptive adjectives. A total mood disturbance (TMD) score is computed from adding all subscales. High scores reflect high mood disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Fadel Zeidan, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arsenault M, Ladouceur A, Lehmann A, Rainville P, Piche M. Pain modulation induced by respiration: phase and frequency effects. Neuroscience. 2013 Nov 12;252:501-11. doi: 10.1016/j.neuroscience.2013.07.048. Epub 2013 Jul 29. PMID 23906637
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Borkovec TD, & Nau, S.D. Credibility of analogue therapy rationales. Journal of Behavior Therapy and Experimental Psychiatry 1972;3:257-260.
- [Background] Buhle J, Wager TD. Does meditation training lead to enduring changes in the anticipation and experience of pain? Pain. 2010 Sep;150(3):382-383. doi: 10.1016/j.pain.2010.05.004. Epub 2010 May 23. No abstract available. PMID 20546996
- [Background] Cassidy EL, Atherton RJ, Robertson N, Walsh DA, Gillett R. Mindfulness, functioning and catastrophizing after multidisciplinary pain management for chronic low back pain. Pain. 2012 Mar;153(3):644-650. doi: 10.1016/j.pain.2011.11.027. Epub 2012 Jan 11. PMID 22240149
- [Background] Coghill RC, Eisenach J. Individual differences in pain sensitivity: implications for treatment decisions. Anesthesiology. 2003 Jun;98(6):1312-4. doi: 10.1097/00000542-200306000-00003. No abstract available. PMID 12766637
- [Background] Coghill RC, Gilron I, Iadarola MJ. Hemispheric lateralization of somatosensory processing. J Neurophysiol. 2001 Jun;85(6):2602-12. doi: 10.1152/jn.2001.85.6.2602. PMID 11387404
- [Background] Coghill RC, Mayer DJ, Price DD. The roles of spatial recruitment and discharge frequency in spinal cord coding of pain: a combined electrophysiological and imaging investigation. Pain. 1993 Jun;53(3):295-309. doi: 10.1016/0304-3959(93)90226-F. PMID 8351159
- [Background] Coghill RC, McHaffie JG, Yen YF. Neural correlates of interindividual differences in the subjective experience of pain. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8538-42. doi: 10.1073/pnas.1430684100. Epub 2003 Jun 24. PMID 12824463
- [Background] Coghill RC, Sang CN, Berman KF, Bennett GJ, Iadarola MJ. Global cerebral blood flow decreases during pain. J Cereb Blood Flow Metab. 1998 Feb;18(2):141-7. doi: 10.1097/00004647-199802000-00003. PMID 9469155
- [Background] Day MA, Smitherman A, Ward LC, Thorn BE. An investigation of the associations between measures of mindfulness and pain catastrophizing. Clin J Pain. 2015 Mar;31(3):222-8. doi: 10.1097/AJP.0000000000000102. PMID 24699159
- [Background] de Boer MJ, Steinhagen HE, Versteegen GJ, Struys MM, Sanderman R. Mindfulness, acceptance and catastrophizing in chronic pain. PLoS One. 2014 Jan 29;9(1):e87445. doi: 10.1371/journal.pone.0087445. eCollection 2014. PMID 24489915
- [Background] Friston KJ, Buechel C, Fink GR, Morris J, Rolls E, Dolan RJ. Psychophysiological and modulatory interactions in neuroimaging. Neuroimage. 1997 Oct;6(3):218-29. doi: 10.1006/nimg.1997.0291. PMID 9344826
- [Background] Gard T, Holzel BK, Sack AT, Hempel H, Lazar SW, Vaitl D, Ott U. Pain attenuation through mindfulness is associated with decreased cognitive control and increased sensory processing in the brain. Cereb Cortex. 2012 Nov;22(11):2692-702. doi: 10.1093/cercor/bhr352. Epub 2011 Dec 15. PMID 22172578
- [Background] Garland EL, Gaylord SA, Palsson O, Faurot K, Douglas Mann J, Whitehead WE. Therapeutic mechanisms of a mindfulness-based treatment for IBS: effects on visceral sensitivity, catastrophizing, and affective processing of pain sensations. J Behav Med. 2012 Dec;35(6):591-602. doi: 10.1007/s10865-011-9391-z. Epub 2011 Dec 8. PMID 22161025
- [Background] Grant JA, Courtemanche J, Duerden EG, Duncan GH, Rainville P. Cortical thickness and pain sensitivity in zen meditators. Emotion. 2010 Feb;10(1):43-53. doi: 10.1037/a0018334. PMID 20141301
- [Background] Grant JA, Rainville P. Pain sensitivity and analgesic effects of mindful states in Zen meditators: a cross-sectional study. Psychosom Med. 2009 Jan;71(1):106-14. doi: 10.1097/PSY.0b013e31818f52ee. Epub 2008 Dec 10. PMID 19073756
- [Background] Jermann F, Billieux J, Laroi F, d'Argembeau A, Bondolfi G, Zermatten A, Van der Linden M. Mindful Attention Awareness Scale (MAAS): Psychometric properties of the French translation and exploration of its relations with emotion regulation strategies. Psychol Assess. 2009 Dec;21(4):506-14. doi: 10.1037/a0017032. PMID 19947785
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Kotov R, Bellman, S., & Watson, D. Multidimensional Iowa suggestibility scale: Brief Manual, 2007.
- [Background] Koyama T, McHaffie JG, Laurienti PJ, Coghill RC. The subjective experience of pain: where expectations become reality. Proc Natl Acad Sci U S A. 2005 Sep 6;102(36):12950-5. doi: 10.1073/pnas.0408576102. Epub 2005 Sep 6. PMID 16150703
- [Background] Lazar SW, Bush G, Gollub RL, Fricchione GL, Khalsa G, Benson H. Functional brain mapping of the relaxation response and meditation. Neuroreport. 2000 May 15;11(7):1581-5. PMID 10841380
- [Background] Lutz A, Greischar LL, Perlman DM, Davidson RJ. BOLD signal in insula is differentially related to cardiac function during compassion meditation in experts vs. novices. Neuroimage. 2009 Sep;47(3):1038-46. doi: 10.1016/j.neuroimage.2009.04.081. Epub 2009 May 5. PMID 19426817
- [Background] McNAir D, Loor, M., & Droppleman, L. Profile of Mood States. San Diego, CA: Educational and Industrial Testing Service, 1971.
- [Background] O'Grady KE. The Absorption Scale: a factor-analytic assessment. Int J Clin Exp Hypn. 1980 Jul;28(3):281-8. doi: 10.1080/00207148008409853. No abstract available. PMID 7390668
- [Background] O'Reilly JX, Woolrich MW, Behrens TE, Smith SM, Johansen-Berg H. Tools of the trade: psychophysiological interactions and functional connectivity. Soc Cogn Affect Neurosci. 2012 Jun;7(5):604-9. doi: 10.1093/scan/nss055. Epub 2012 May 7. PMID 22569188
- [Background] Perlman DM, Salomons TV, Davidson RJ, Lutz A. Differential effects on pain intensity and unpleasantness of two meditation practices. Emotion. 2010 Feb;10(1):65-71. doi: 10.1037/a0018440. PMID 20141303
- [Background] Petrovic P, Kalso E, Petersson KM, Andersson J, Fransson P, Ingvar M. A prefrontal non-opioid mechanism in placebo analgesia. Pain. 2010 Jul;150(1):59-65. doi: 10.1016/j.pain.2010.03.011. PMID 20399560
- [Background] Peyron R, Garcia-Larrea L, Gregoire MC, Convers P, Richard A, Lavenne F, Barral FG, Mauguiere F, Michel D, Laurent B. Parietal and cingulate processes in central pain. A combined positron emission tomography (PET) and functional magnetic resonance imaging (fMRI) study of an unusual case. Pain. 2000 Jan;84(1):77-87. doi: 10.1016/S0304-3959(99)00190-6. PMID 10601675
- [Background] Poulin PA, Romanow HC, Rahbari N, Small R, Smyth CE, Hatchard T, Solomon BK, Song X, Harris CA, Kowal J, Nathan HJ, Wilson KG. The relationship between mindfulness, pain intensity, pain catastrophizing, depression, and quality of life among cancer survivors living with chronic neuropathic pain. Support Care Cancer. 2016 Oct;24(10):4167-75. doi: 10.1007/s00520-016-3243-x. Epub 2016 May 18. PMID 27193116
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Price DD, Harkins SW, Baker C. Sensory-affective relationships among different types of clinical and experimental pain. Pain. 1987 Mar;28(3):297-307. doi: 10.1016/0304-3959(87)90065-0. PMID 2952934
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Prins B, Decuypere A, Van Damme S. Effects of mindfulness and distraction on pain depend upon individual differences in pain catastrophizing: an experimental study. Eur J Pain. 2014 Oct;18(9):1307-15. doi: 10.1002/j.1532-2149.2014.491.x. Epub 2014 Mar 26. PMID 24677437
- [Background] Rainville P, Duncan GH, Price DD, Carrier B, Bushnell MC. Pain affect encoded in human anterior cingulate but not somatosensory cortex. Science. 1997 Aug 15;277(5328):968-71. doi: 10.1126/science.277.5328.968. PMID 9252330
- [Background] Rhudy JL. Respiration-induced hypoalgesia: additional evidence for pain modulation deficits in fibromyalgia? Pain. 2010 Apr;149(1):1-2. doi: 10.1016/j.pain.2010.01.004. Epub 2010 Feb 1. No abstract available. PMID 20122804
- [Background] Salkind MR. Beck depression inventory in general practice. J R Coll Gen Pract. 1969 Nov;18(88):267-71. No abstract available. PMID 5350525
- [Background] Schutze R, Rees C, Preece M, Schutze M. Low mindfulness predicts pain catastrophizing in a fear-avoidance model of chronic pain. Pain. 2010 Jan;148(1):120-127. doi: 10.1016/j.pain.2009.10.030. Epub 2009 Nov 26. PMID 19944534
- [Background] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory (STAI-form y). Palo Alto, CA: Consulting Psychology Press, 1983.
- [Background] Starr CJ, Sawaki L, Wittenberg GF, Burdette JH, Oshiro Y, Quevedo AS, Coghill RC. Roles of the insular cortex in the modulation of pain: insights from brain lesions. J Neurosci. 2009 Mar 4;29(9):2684-94. doi: 10.1523/JNEUROSCI.5173-08.2009. PMID 19261863
- [Background] Sullivan MJ, D'Eon JL. Relation between catastrophizing and depression in chronic pain patients. J Abnorm Psychol. 1990 Aug;99(3):260-3. doi: 10.1037//0021-843x.99.3.260. PMID 2145334
- [Background] Sullivan MJL, Martel MO, Tripp D, Savard A, Crombez G. The relation between catastrophizing and the communication of pain experience. Pain. 2006 Jun;122(3):282-288. doi: 10.1016/j.pain.2006.02.001. Epub 2006 Mar 20. PMID 16545907
- [Background] Sullivan MJL, Stanish W, Waite H, Sullivan M, Tripp DA. Catastrophizing, pain, and disability in patients with soft-tissue injuries. Pain. 1998 Sep;77(3):253-260. doi: 10.1016/S0304-3959(98)00097-9. PMID 9808350
- [Background] Tang YY, Ma Y, Wang J, Fan Y, Feng S, Lu Q, Yu Q, Sui D, Rothbart MK, Fan M, Posner MI. Short-term meditation training improves attention and self-regulation. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17152-6. doi: 10.1073/pnas.0707678104. Epub 2007 Oct 11. PMID 17940025
- [Background] Velanovich V, Younga J, Bhandarkar V, Marshall N, McLaren P, Ritz J, Rubinfeld I. A single, global patient-centered measure from the SF-36 instrument to assess surgical outcomes and quality of life: a pilot study. World J Surg. 2012 Sep;36(9):2045-50. doi: 10.1007/s00268-012-1634-9. PMID 22538393
- [Background] Villemure C, Bushnell MC. Mood influences supraspinal pain processing separately from attention. J Neurosci. 2009 Jan 21;29(3):705-15. doi: 10.1523/JNEUROSCI.3822-08.2009. PMID 19158297
- [Background] Wager TD, Rilling JK, Smith EE, Sokolik A, Casey KL, Davidson RJ, Kosslyn SM, Rose RM, Cohen JD. Placebo-induced changes in FMRI in the anticipation and experience of pain. Science. 2004 Feb 20;303(5661):1162-7. doi: 10.1126/science.1093065. PMID 14976306
- [Background] Walach H, Buchheld N, Buttenmuller V, Kleinknecht N, Schmidt S. Measuring mindfulness-the Freiburg Mindfulness Inventory (FMI). Personality and Individual Differences 2006;40:1543-1555.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] White G. Natural History and Antiquities of Selborne. London, England: Cassell and Company, 1908.
- [Background] Woolrich MW, Ripley BD, Brady M, Smith SM. Temporal autocorrelation in univariate linear modeling of FMRI data. Neuroimage. 2001 Dec;14(6):1370-86. doi: 10.1006/nimg.2001.0931. PMID 11707093
- [Background] Worsley KJ, Evans AC, Marrett S, Neelin P. A three-dimensional statistical analysis for CBF activation studies in human brain. J Cereb Blood Flow Metab. 1992 Nov;12(6):900-18. doi: 10.1038/jcbfm.1992.127. PMID 1400644
- [Background] Yelle MD, Oshiro Y, Kraft RA, Coghill RC. Temporal filtering of nociceptive information by dynamic activation of endogenous pain modulatory systems. J Neurosci. 2009 Aug 19;29(33):10264-71. doi: 10.1523/JNEUROSCI.4648-08.2009. PMID 19692600
- [Background] Zeidan F. The Neurobiology of Mindfulness Meditation. In: KW Brown, Creswell, J.D., & R.M., Ryan, editor. Handbook of Mindfulness Science: Theory, Research and Practice. New York, New York: The Guilford Press, 2015.
- [Background] Zeidan F, Adler-Neal AL, Wells RE, Stagnaro E, May LM, Eisenach JC, McHaffie JG, Coghill RC. Mindfulness-Meditation-Based Pain Relief Is Not Mediated by Endogenous Opioids. J Neurosci. 2016 Mar 16;36(11):3391-7. doi: 10.1523/JNEUROSCI.4328-15.2016. PMID 26985045
- [Background] Zeidan F, Emerson NM, Farris SR, Ray JN, Jung Y, McHaffie JG, Coghill RC. Mindfulness Meditation-Based Pain Relief Employs Different Neural Mechanisms Than Placebo and Sham Mindfulness Meditation-Induced Analgesia. J Neurosci. 2015 Nov 18;35(46):15307-25. doi: 10.1523/JNEUROSCI.2542-15.2015. PMID 26586819
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Zeidan F, Grant JA, Brown CA, McHaffie JG, Coghill RC. Mindfulness meditation-related pain relief: evidence for unique brain mechanisms in the regulation of pain. Neurosci Lett. 2012 Jun 29;520(2):165-73. doi: 10.1016/j.neulet.2012.03.082. Epub 2012 Apr 6. PMID 22487846
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Zeidan F, Johnson SK, Gordon NS, Goolkasian P. Effects of brief and sham mindfulness meditation on mood and cardiovascular variables. J Altern Complement Med. 2010 Aug;16(8):867-73. doi: 10.1089/acm.2009.0321. PMID 20666590
- [Background] Zeidan F, Lobanov OV, Kraft RA, Coghill RC. Brain mechanisms supporting violated expectations of pain. Pain. 2015 Sep;156(9):1772-1785. doi: 10.1097/j.pain.0000000000000231. PMID 26083664
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390